CLINICAL TRIAL: NCT01376414
Title: Pilot Study to Estimate the Prevalence of Helicobacter Pylori (H. Pylori) Infection in Patients Presenting With Non-specific Upper Abdominal Pain to the Emergency Department (ED.)
Brief Title: H. Pylori Testing for Patients With Non-specific Upper Abdominal Pain in the Emergency Department
Status: Completed | Type: Observational
Sponsor: George Washington University (Other)
Responsible Party: Sponsor
Other Study IDs: IRB#: 111050
Record Dates: First submitted 2011-06-16; First posted 2011-06-20 (Estimated); Last update posted 2016-08-26 (Estimated); Status verified 2012-08

CONDITIONS: Gastritis; Peptic Ulcer; Peptic Ulcer Perforation; Stomach Ulcer
Keywords: dyspepsia; abdominal; pain; helicobacter; pylori; [C06.405.748.398]; [C06.405.748.586]; [C06.405.748.586.698]; [C06.405.748.586.849]
MeSH Terms: conditions — Gastritis; Peptic Ulcer; Peptic Ulcer Perforation; Stomach Ulcer; Dyspepsia; Pain | interventions — Emergency Service, Hospital

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Non specific upper abdominal pain: Cohort is patients who present to the Emergency Department with primary complaint of upper abdominal pain without obvious cause.
  Interventions: Other: Urea Breath Test (UBT) for H. pylori infection

INTERVENTIONS:
Other: Urea Breath Test (UBT) for H. pylori infection — 13C UBT to detect H. pylori infection. Single bedside test that determines infection in about ten minutes. Test machine is a product of Exalenz bioscience.
  Other Names: 13C; UBT; H. pylori; helicobacter; gastric; ulcers; dyspepsia; emergency; abdominal pain; exalenz

SUMMARY:
This pilot study aims to estimate the prevalence of Helicobacter pylori (H. pylori) colonization in patients presenting with non-specific abdominal pain (NSAP) in an urban academic emergency department (ED) located in Washington, DC.

DETAILED DESCRIPTION:
The major goal is to study the prevalence of H. pylori using the 13C Urea Breath Test (UBT) in emergency department (ED) patients with non-specific abdominal pain. The investigators plan to enroll 250 patients during the pilot stage of this study. This T2 translational trial aims to apply recommended guidelines for the investigation and management of NSAP and dyspepsia into the practical arena of ED clinical care. The "test-and-treat" approach to symptomatic H. pylori infection has been endorsed by the American Gastroenterological Association (AGA). Patients who test positive for H. pylori by UBT will be treated with clarithromycin-based triple medication therapy as recommended by the American College of Gastroenterology (ACG) at the discretion of the treating physician. The rationale is that successful identification of H. pylori in the ED and initiation of treatment may reduce future risk of gastritis, gastric lymphoma, and gastric cancer, and is cost-effective through reduction of future healthcare costs and symptom severity. Study subjects will be followed for medication compliance, resolution of symptoms, and ability to obtain outpatient follow-up. As part of this study, the investigators will be collecting important information on the ED evaluation of abdominal pain.

ELIGIBILITY:
Inclusion Criteria:

For any patient with chief complaint of "ABD", "STOM", "EPIG", "CHEST", "NAUS" "Do you have pain or discomfort or burning in your upper abdomen as the main reason for coming to ER today?"

Exclusion Criteria:

* The patient LESS than 18 years old.
* Patient does NOT speak English NOR has reliable adult translator.
* Patient does NOT have capacity to give consent? (confused/intoxicated/etc.)
* The patient currently is on antibiotics.
* The patient currently is on a PPI. (eg. Prilosec [omeprazole]), protonix [pantoprazole], prevacid [lansoprazole], aciphex [rabeprazole], nexium [esomeprazole]
* The patient has taken bismuth or pepto-bismol today.
* The patient is known to be or suspected to be pregnant.
* The patient UNABLE to walk to H.pylori Breath test.
* The patient had "recent" negative H.pylori test for same symptoms.
* There an "obvious alternative cause" for pain (per attending).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adult patients (>18 years) presenting to the ED with symptoms of abdominal pain will be screened for eligibility. The ED is a single site urban academic level one trauma center.
Sampling Method: Non-Probability Sample
Enrollment: 212 (Actual)
Dates: Start 2011-03; Primary Completion 2014-08 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Prevalence of H. pylori infection in ED patients with symptomatic abdominal pain | 6 momths
  Prevalence of H. pylori infection diagnosed by UBT in patients with symptomatic upper abdominal pain treated in the ED.

SECONDARY OUTCOMES:
SES measures | 6 months
  DoeS SES correlate with HP infection?

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - George Washington University Hospital, Washington D.C., District of Columbia
  - GWU Hospital, Washington D.C., District of Columbia